CLINICAL TRIAL: NCT05743998
Title: Inactivity and Health Related Quality of Life in Dialysis Patients and Peritoneal Dialysis Patients
Brief Title: Inactivity and Quality of Life in Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Pardis Specialized Wellness Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PA23ES-1-01
Record Dates: First submitted 2023-02-10; First posted 2023-02-24 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Chronic Kidney Diseases; End Stage Renal Disease; Hemodialysis Complication; Peritoneal Dialysis
Keywords: Inactivity; Quality of life; Physical activity; Sedentary lifestyle; Peritoneal Dialysis; Hemodialysis; Exercise
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemodialysis patients: They will fill 2 questionnaires and ill do some functional tests.
- Peritoneal dialysis patients: They will fill 2 questionnaires and ill do some functional tests.

SUMMARY:
The goal of this observational study is to compare hemodialysis and peritoneal dialysis patients. The main questions it mains to answer are:

* What is the level of physical activity in hemodialysis and peritoneal dialysis patients?
* What is the level of quality of life of hemodialysis and peritoneal dialysis patients?
* Is there any relation between inactivity and quality of life in hemodialysis and peritoneal dialysis patients?

Participants will answer 2 questionnaires and will do some functional tests.

DETAILED DESCRIPTION:
Physical functioning and physical activity are low in patients treated with maintenance hemodialysis (HD).

One of the factors that lead to a further decrease in the activity of hemodialysis patients and its complications is the immobility of these patients during hemodialysis. This method of treatment forces patients to remain motionless for 4 hours on average 3 times a week. In addition, fatigue after dialysis also requires additional rest and immobility for about 2 to 6 hours.

Sedentary behaviors are also common in peritoneal dialysis (PD) patients (about 63%), and studies have shown that there is no significant difference between the physical activity level of PD and HD patients.

In PD patients, in addition to reducing functional capacity and feeling extreme fatigue, the fear of dialysis fluid leakage, hernia and infection also causes a decrease in physical activity and an increase in inactivity in these patients.

The lack of physical mobility and the resulting movement restrictions affect the patient's independence and ability to perform daily tasks, including self-care. In addition, the emotional and mental health of patients is greatly affected by these restrictions Inactivity sets off a vicious cycle in which energy imbalances can increase comorbidities such as hypertension, diabetes, coronary artery disease, depressive disorders, hospitalization rates, and disability. Each of these conditions aggravates the decrease in the quality of life and increases the mortality of patients.

Quality of life is an important aspect of treatment outcomes and should be considered when evaluating the quality and effectiveness of renal care services.

The quality of life in CKD patients and especially dialysis patients decreases under the influence of several factors such as weakness, disability, reduced functional capacity, anemia, malnutrition, impaired cognitive function, worsening sleep quality, increased depression, and the development of cardiovascular disorders The quality of life of renal patients and its social and emotional aspects are considered as the main determinants of these clinical outcomes.

Decreasing the quality of life in hemodialysis patients and peritoneal dialysis patients decreases the survival and increases the mortality of these patients. Improving the quality of life should not only be considered as a therapeutic goal in itself, but should also be considered as an essential factor in reducing the number of hospitalizations and deaths of dialysis patients.

This study aims to evaluate the quality of life of HD patients as well as PD patients. Also this study will evaluate the effect of inactivity on quality of life, stratified by both dialysis modality and will compere the results in these two dialysis modalities.

ELIGIBILITY:
Inclusion Criteria:

* being treated with the same respective dialysis modalities for at least 3 months
* being ambulatory (with or without assistive device)
* ability to understand and provide informed consent

Exclusion Criteria:

* non-ambulatory
* had significant cognitive dysfunction
* progressive degenerative
* neurologic disease
* severe rheumatologic or orthopedic conditions that would limit and would be exacerbated by the testing
* angina upon exertion, or myocardial infarction or cardiac surgery within the last year.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis and peritoneal dialysis patients being treated with the same respective dialysis modalities for at least 3 months and being ambulatory (with or without assistive device) will be included.
  But non-ambulatory patients having significant cognitive dysfunction, progressive degenerative,neurologic disease or severe rheumatologic or orthopedic conditions, angina upon exertion, or myocardial infarction or cardiac surgery within the last year will be excluded.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Quality of life level | Through out study completion, an average of 2 weeks
  Quality of life will be assessed by health related quality of life questionnaire for chronic kidney disease patients Higher scores indicate higher levels of quality of life
Physical activity level | Through out study completion, an average of 2 weeks
  Physical activity level will be assessed by Low Physical activity questionnaire (LoPAQ) This questionnaire assesses the levels of physical activity and will be explained by calories expenditure. Those who are less active will have lower calories expenditure.

SECONDARY OUTCOMES:
Physical functioning level | Through out study completion, an average of 2 weeks
  Physical functioning level will be assessed by short physical performance battery test.
  The range of this test score is 0-12. Those who have disabilities in the activity of their daily living will take lower scores.

CONTACTS AND LOCATIONS:
Overall Officials: MohammadAli Tabibi, PhD, Principal Investigator — Pardis Specialized Wellness Institute
Locations (1):
- Khorshid Dialysis Center, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published article, after deidentification are to be shared.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available after the paper is published. No end date.
Access Criteria: Data will be accessible with no criteria. Anyone who wishes will have access to data.

REFERENCES:
- [Result] Ramer SJ, McCall NN, Robinson-Cohen C, Siew ED, Salat H, Bian A, Stewart TG, El-Sourady MH, Karlekar M, Lipworth L, Ikizler TA, Abdel-Kader K. Health Outcome Priorities of Older Adults with Advanced CKD and Concordance with Their Nephrology Providers' Perceptions. J Am Soc Nephrol. 2018 Dec;29(12):2870-2878. doi: 10.1681/ASN.2018060657. Epub 2018 Nov 1. PMID 30385652
- [Result] DeOreo PB. Hemodialysis patient-assessed functional health status predicts continued survival, hospitalization, and dialysis-attendance compliance. Am J Kidney Dis. 1997 Aug;30(2):204-12. doi: 10.1016/s0272-6386(97)90053-6. PMID 9261030
- [Result] Painter P, Roshanravan B. The association of physical activity and physical function with clinical outcomes in adults with chronic kidney disease. Curr Opin Nephrol Hypertens. 2013 Nov;22(6):615-23. doi: 10.1097/MNH.0b013e328365b43a. PMID 24100215
- [Result] Luk WS. Rehabilitation services for patients undergoing peritoneal dialysis in Hong Kong. Nurs Stand. 2006 Jan 25-31;20(20):41-7. doi: 10.7748/ns2006.01.20.20.41.c4049. PMID 16459764
- [Result] Ulutas O, Farragher J, Chiu E, Cook WL, Jassal SV. Functional Disability in Older Adults Maintained on Peritoneal Dialysis Therapy. Perit Dial Int. 2016 Jan-Feb;36(1):71-8. doi: 10.3747/pdi.2013.00293. Epub 2014 Apr 7. PMID 24711642
- [Result] Roshanravan B, Robinson-Cohen C, Patel KV, Ayers E, Littman AJ, de Boer IH, Ikizler TA, Himmelfarb J, Katzel LI, Kestenbaum B, Seliger S. Association between physical performance and all-cause mortality in CKD. J Am Soc Nephrol. 2013 Apr;24(5):822-30. doi: 10.1681/ASN.2012070702. Epub 2013 Apr 18. PMID 23599380